CLINICAL TRIAL: NCT04483154
Title: Perry Virtual - A Prospective and Observational Rural Health Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Coala Life, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: #20-PCHO-101
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: COPD; Arrhythmia; Murmur, Heart; Chronic Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Arrhythmias, Cardiac; Heart Murmurs; Chronic Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Coala Heart Monitor — The Coala Heart Monitor (Coala Life AB, Sweden) is a CE and FDA-cleared device for real-time, remote monitoring of 2-lead ECG as well as heart and lung sounds. The Coala Heart Monitor automatically detects for 9 of the most common arrhythmias and has an integrated stethoscope for remote auscultation. It is paired wirelessly with the patient's smartphone and results are provided instantly both to patient and to connected provider in the cloud-based Coala Care portal.

SUMMARY:
The principal objective of the study is to determine if patient-empowered, real-time and home- based patient monitoring of vital parameters can lead to:

* Reduction in admission rates and improved clinical management of chronically ill patients
* Reduction in use of medications
* Reported quality of life

A minimum of 100 patients will be recruited, monitored and observed over 6 months from home with the Coala Heart Monitor. The study population will be representative of rural, high-risk, Medicare (65+ of age) subjects with chronic conditions and will be recruited by the Perry Community Hospital in Linden, TN.

DETAILED DESCRIPTION:
More than 46 million Americans, or 15% of the US population, live in rural areas. According to the Center of Disease Control (CDC), rural Americans face numerous health disparities and more likely to die from heart disease, cancer, unintentional injury, chronic lower respiratory disease, and stroke than their urban counterparts. A series of studies from CDC have drawn attention to the significant gap in health between rural and urban Americans.

Heart palpitations account for over 70 million US primary care visits every year and is the second most common reason for visiting a cardiologist in the US. With the increased availability of single-lead consumer ECG solutions increasing the demand on providers, home- based solutions are needed enabling cost-effective, prescription-based and diagnostic monitoring solution are needed.

The Coala Heart Monitor was introduced in Scandinavia in 2017 and in the US in 2019. The device is connected to the patient's smartphone and records ECG as well as heart and lung sounds.The complementary cloud-based data analytics platform, Coala Care, analyzes the full disclosed, high resolution data using smart algorithms to detect cardiac rhythm deviations by advanced pattern recognition including real-time AFib detection based on P-waves and R-R dispersion. The heart sounds are further transformed into high-fidelity phonocardiograms (PCG) for murmur detection in real time. Heart and lung sounds can be listened to remotely.

Both health care providers and patients can view the results - the former via the HIPAA- compliant online portal and the latter via the Coala smartphone app - and physicians can send secure private messages immediately if something requires a follow-up.

The COVID-19 Coronavirus pandemic has quickly transformed cardiovascular medicine with shift from traditional hands-on care to remote hands-off telemedicine to keep patients and their medical staff safe.

ELIGIBILITY:
Inclusion Criteria:

* History of frequent admissions, defined as minimum of 2 during the last 6 months
* ICD diagnosis for COPD and/or hypertension and/or diabetes and/or cardiovascular diseases
* Patient has Smartphone or Tablet, as well as Internet connection in their homes (or 3G/4G/5G connection)

Exclusion Criteria:

* Subjects with Pacemaker, ICD or Implanted Loop Recorder
* Subjects with no experience in using Smartphones and Apps
* Vulnerable Subjects (prisoners, elderly with decisional incapacity)

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Rural population with chronic illnesses and high admission rates
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Reducing admission rates | 6 months
Reduction in use of medications | 6 months
Increased quality of life | 6 months
  As measured by Rand-36
Improved clinical management | 6 months

SECONDARY OUTCOMES:
Show the value of using Coala Heart Monitor in rural care - patients | 6 months
Show the value of using Coala Heart Monitor in rural care - providers | 6 months
  The cloud-based Coala Care platform enables patient data to be shared and accessed efficiently with affiliated specialists. Show how this helps improve clinical management and healthcare processes.

CONTACTS AND LOCATIONS:
Overall Officials: David Huneycutt, MD, Principal Investigator — Perry Community Hospital
Locations (1):
- Perry Community Hospital, Linden, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided